CLINICAL TRIAL: NCT03883100
Title: A Phase II Multi-center, Open Label Study of HQP1351 in Chinese Patients of Chronic Myeloid Leukemia With T315I Mutation in Accelerated Phase
Brief Title: A Pivotal Study of HQP1351 in Patients of Chronic Myeloid Leukemia in Accelerated Phase With T315I Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HQP1351CC202
Record Dates: First submitted 2019-03-13; First posted 2019-03-20 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Chronic Myeloid Leukemia - Accelerated Phase
Keywords: Chronic Myeloid Leukemia,CML; T315I mutation; CML-AP; HQP1351; Olverembatinib Tablets
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase | interventions — olverembatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HQP1351 (Experimental)
  Interventions: Drug: HQP1351

INTERVENTIONS:
Drug: HQP1351 — 40 mg tablet, taken orally once every other day

SUMMARY:
The purpose of this study is to evaluate the efficacy of HQP1351 in patients with chronic myeloid leukemia in accelerated phase (CML-AP) harboring T315I mutation. The efficacy of HQP1351 was determined by evaluating the subjects' major hematologic response (MaHR).

DETAILED DESCRIPTION:
This is an open, single-arm, multi-center phase 2 clinical study to evaluate the efficacy and safety of oral administrated of HQP1351(40mg, QOD) in CML-AP patients with T315I mutation in China. A total of 20 CML-AP patients will be included in this pivotal study. After screening, eligible subjects will receive oral HQP1351 40mg on a continues once every other day dosing regimen, until disease progression, drug intolerance, or meet other treatment conditions to discontinue the study. During the course of treatment, each subject will be assessed regularly for hematological, cytogenetic and molecular responses. At the same time, safety information also will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female patients who are 18 years of age or older.
2. CML-AP patients with positive Ph chromosome or BCR-ABL fusion genes.
3. After any targeted BCR-ABL1 tyrosine kinase inhibitors (TKI) treatment, CML-AP patients with T315I mutation.
4. Ability to understand and willingness to sign a written informed consent form. The consent form must be signed by the patient prior to any study-specific procedures.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
6. Predicted life expectancy of ≥3 months.
7. Organ function as indicated by the following laboratory indicators must be met（Hematological indicators require that no blood transfusion or any blood products or cytokines be used within 14 days prior to testing）:

   * Hemoglobin ≥8.0g/dL.
   * White blood cell count ≥ 3.0×10^9/L.
   * Platelet count ≥ 75×10^9/L.
   * Serum creatinine ≤ 1.5×upper limit of normal (ULN) or 24 hours calculated creatinine clearance ≥ 50mL/min when serum creatinine >1.5×ULN.
   * Serum albumin ≥ 3.0 g/dL.
   * Total bilirubin ≤ 1.5 x ULN.
   * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x ULN.
   * Amylase≤1.5×ULN. Lipase≤1.5×ULN.
   * PT、APTT、INR≤1.5×ULN.
8. Cardiac function index: ejection fraction (EF) > 50%, pulmonary arterial systolic pressure (PASP) ≤50 mmHg.
9. QT interval corrected on electrocardiogram (ECG) evaluation: QTc≤450ms in males or ≤470ms in females.
10. Males and females of childbearing potential and their partners voluntarily take contraceptive measures that the researchers believe are effective within 120 days from the signing of the informed consent to the last use of the research drug, or confirm that sterilization has been performed (at least one month before screening).
11. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

1. Received cytotoxic chemotherapy or radiotherapy within 28 days prior to the first administration, interferon or cytarabine or antitumor effect Chinese herbal medicine or Chinese patent medicine within 14 days prior to the first administration, or targeted BCR-ABL1 TKI within 7 days prior to the first administration, or hydroxyurea or anagrelide within 24 hours after the first administration, or adverse events (except alopecia) caused by previous treatment and have not recovered.
2. The patients who received any other investigating drugs within 14 days prior to first administration.
3. Patients who have progressed to blast phase (BP) in the past.
4. Patients who are currently receiving treatment with a medication that has the potential to interact with research drug.
5. Have previously been treated with ponatinib or HQP1351 (or drugs of similar composition).
6. Absorption disorder syndrome or other diseases affecting oral drug absorption.
7. Have any history of heart or vascular disease, such as hypertension (systolic blood pressure(HBP) > 140mmHg and/or diastolic blood pressure > 90mmHg), or take medications that are known to cause QT interval prolongation. The patients with well controlled HBP can be considered to be included.
8. Pulmonary systolic pressure (PSP) of echocardiography is more than 50 mmHg, or there is clinical symptom related to pulmonary hypertension.
9. Have a history of serious cardiovascular diseases during the previous treatment of chronic myeloid leukemia with TKI, including myocardial infarction, unstable angina pectoris, severe arrhythmia and congestive heart failure.
10. Underwent autologous or allogeneic stem cell transplant.
11. CML-AP patient currently diagnosed as major hematologic response (MaHR).
12. Have diseases with abnormal bleeding and coagulation function, or have a bleeding disorder unrelated to CML within 3 months before first dose of study drug.
13. Underwent major surgery (except minor surgical procedures, such as placement or bone marrow biopsy) with 14 days prior to the first dose of study drug.
14. Require concurrent treatment with immunosuppressive agents, other than corticosteroids prescribed for a short course of therapy (It is defined as a daily dose of corticosteroids less than 30 mg prednisone or the same amount of other corticosteroids within 7 days).
15. Have active nervous system (CNS) disease as evidence by cytology or pathology. In the absence of clinical CNS disease, lumbar puncture is not required.
16. History of another primary malignancies.
17. Active symptomatic infection.
18. Known to be allergic to study drug ingredients or their analogues.
19. Female patients with blood β-Human chorionic gonadotropin positive, pregnant or lactating or expecting pregnancy during the study program.
20. Suffer from any condition or illness that, in the opinion of the Investigator, would compromise patient safety or interfere with the evaluation of the safety of the research drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Major hematologic response (MaHR) | By the end of Cycle 24 (each cycle is 28 days)
  MaHR is the proportion of patients achieving Complete hematologic response (CHR) or no evidence of leukemia (NEL). It is defined as the best response obtained by the subjects during the whole treatment process of the study.

SECONDARY OUTCOMES:
CHR | By the end of Cycle 24 (each cycle is 28 days)
  CHR is the proportion of patients achieving CHR after being treated with HQP1351. It is defined as the best response obtained by the subjects during the whole treatment process of the study.
Major cytogenetic response (MCyR) | By the end of Cycle 24 (each cycle is 28 days)
  MCyR is the proportion of patients achieving Complete cytogenetic response (CCyR: defined as 0% Philadelphia chromosome-positive [Ph+] metaphases by cytogenetic analysis of bone marrow) or Partial Cytogenetic Response (PCyR: defined as >0% to 35% Ph+ metaphases by cytogenetic analysis of bone marrow). It is defined as the best response obtained by the subjects during the whole treatment process of the study.
CCyR | By the end of Cycle 24 (each cycle is 28 days)
  CCyR is the proportion of patients achieving CCyR after being treated with HQP1351. It is defined as the best response obtained by the subjects during the whole treatment process of the study.
Major molecular response (MMR) | By the end of Cycle 24 (each cycle is 28 days)
  MMR is the proportion of patients achieving a ratio of ≤0.1% breakpoint cluster region (BCR) abelson leukemia (ABL) to ABL transcripts on the international scale (≤0.1% BCR-ABL/ABL[IS]) after being treated with HQP1351. It is defined as the best response obtained by the subjects during the whole treatment process of the study.
Time to response | By the end of Cycle 24 (each cycle is 28 days)
  The time to response is defined as the interval between the first use of HQP1351 and the first date at which the criteria for response are met. The subject who isn't met the response criteria will be censored at the last assessment time.
Duration of response | By the end of Cycle 24 (each cycle is 28 days)
  Duration of response is defined as the interval between the first assessment at which the criteria for response are met until the earliest date at which the criteria for progression are met, and the subject who isn't met the progression criteria will be censored at the last assessment time. The duration of response is calculated only for subjects who achieved response.
Progression free survival (PFS) | By the end of Cycle 24 (each cycle is 28 days)
  PFS is defined as the interval between the first dose date of HQP1351 treatment and the first date at which the criteria for progression are met, or death. The subject who isn't progression or death will be censored at the last response assessment.
Overall survive (OS) | By the end of Cycle 24 (each cycle is 28 days)
  OS is defined as the interval between the first dose date of HQP1351 treatment and date of death, censored at the last contact date to be alive.
Safety: adverse events (AEs), and serious AEs (SAEs) | By the end of Cycle 24 (each cycle is 28 days)
  Patients with HQP1351 treatment related AE, SAE will be assessed according NCI CTCAE Version 5.0.

OTHER OUTCOMES:
The relationship between mutation and efficacy. | By the end of Cycle 24 (each cycle is 28 days)
  During the course of HQP1351 therapy, the relationship between BCR-ABL1 kinase region/other mutations and drug resistance/disease progression will be measured.
Quality of life (QOL) | By the end of Cycle 24 (each cycle is 28 days)
  Objects' quality of life will be measured during the course of HQP1351 therapy by European Organization for Research and Treatment (EORTC) quality of life questionnaire core-30 version3 [QLQ-C30(V3) questionnaire].

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, Professor, Principal Investigator — Peking University People's Hospital; Qian Jiang, Professor, Principal Investigator — Peking University People's Hospital
Locations (9):
- China (9):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guandong
  - Nanfang hospital of southern medical university, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Henan Tumor Hospital, Zhengzhou, Henan
  - Tongji medical college Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital medical college Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Hospital Affiliated of Soochow University, Suzhou, Jiangsu
  - Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Jiang Q, Li Z, Qin Y, Li W, Xu N, Liu B, Zhang Y, Meng L, Zhu H, Du X, Chen S, Liang Y, Hu Y, Liu X, Song Y, Men L, Chen Z, Niu Q, Wang H, Lu M, Yang D, Zhai Y, Huang X. Olverembatinib (HQP1351), a well-tolerated and effective tyrosine kinase inhibitor for patients with T315I-mutated chronic myeloid leukemia: results of an open-label, multicenter phase 1/2 trial. J Hematol Oncol. 2022 Aug 18;15(1):113. doi: 10.1186/s13045-022-01334-z. PMID 35982483